CLINICAL TRIAL: NCT01038284
Title: Evaluation of Multidisciplinary Collaboration Care Program in Pulmonary Arterial Hypertension
Brief Title: Multidisciplinary Collaboration Care in Pulmonary Arterial Hypertension (PAH)
Acronym: ETHAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: DCIC 09 12
Record Dates: First submitted 2009-10-22; First posted 2009-12-23 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Hypertension, Pulmonary
Keywords: Patient Education; Drug Toxicity
MeSH Terms: conditions — Hypertension, Pulmonary; Drug-Related Side Effects and Adverse Reactions | interventions — Patient Education as Topic; Data Collection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Sham Comparator)
  Interventions: Other: Data collection
- Patient education (Active Comparator)
  Interventions: Behavioral: Patient education

INTERVENTIONS:
Behavioral: Patient education — Pharmaceutical care of patients with PAH
  Arms: Patient education
Other: Data collection — Clinical and biological data, treatment, medication errors and ADEs
  Arms: Control

SUMMARY:
Pulmonary arterial hypertension (PAH) is a severe pulmonary vascular affection, which treatment has evolved in the last few years, improving quality of life. However, adherence to treatment has not been assessed in such patients. The investigators developed a collaborative care model involving clinical pharmacists in PAH. The objective of this work is to evaluate the impact of such model of care on medication errors and adverse events, quality of life and clinical criteria.

This randomized multicentre controlled study will include approximately 100 PAH patients (NYHA II to IV). After inclusion, patients will receive either collaborative care including consultations with specialized pharmacist and nurse, or classic follow-up. Each patient will be followed during 18 months from the date of inclusion.

The investigators hope to show the positive impact of a collaborative care model in PAH. More specifically, the investigators aim to show the interest of long-term patient education to improve patient safety related to drugs, but also their quality of life, and have preliminary data about usual clinical criteria.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18;
* Pulmonary arterial hypertension (NYHA II to IV);
* Any specific PAH treatment or oral anticoagulant.

Exclusion Criteria:

* Patients under 18 or protected by law;
* Patients who do not speak/understand French;
* Pregnancy;
* Patients enrolled in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2010-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Medication-related problems | 18 months
  Medication errors (assessed by using the tool developped by the French Society for Clinical Pharmacy) and adverse drug reactions

SECONDARY OUTCOMES:
Patient Satisfaction with medication | 18 months
  Comparison between the SATMED-Q(R) score at 18 months between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Roustit, PharmD, Study Director — Clinical Research Center - Inserm CIC03, Grenoble, France; Pison Christophe, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (11):
- France (11):
  - CHU Bordeaux, Bordeaux
  - CHU Brest, Brest
  - Hopital Antoine Beclere, Clamart
  - Clinical Research Center Inserm CIC03 - Grenoble University Hospital, Grenoble
  - CHU Grenoble, Grenoble
  - CHU de Lille, Lille
  - CHU Nantes, Nantes
  - CHU de Nice, Nice
  - CHU Rouen, Rouen
  - CHU Strasbourg, Strasbourg
  - CHU Tours, Tours

REFERENCES:
- [Derived] Roustit M, Chaumais MC, Chapuis C, Gairard-Dory A, Hadjadj C, Chanoine S, Allenet B, Sitbon O, Pison C, Bedouch P; ETHAP Study Group. Evaluation of a collaborative care program for pulmonary hypertension patients: a multicenter randomized trial. Int J Clin Pharm. 2020 Aug;42(4):1128-1138. doi: 10.1007/s11096-020-01047-8. Epub 2020 May 21. PMID 32440738